CLINICAL TRIAL: NCT03842202
Title: Effect of Semaglutide 2.4 mg Once-weekly on Gastric Emptying in Subjects With Obesity
Brief Title: A Research Study to Look at How Semaglutide Affects Gastric Emptying in People With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4455; U1111-1215-9915 (Other: World Health Organization (WHO)); 2018-002497-42 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Participants will receive increasing doses of semaglutide. The treatment period from first treatment (Day 1) to end of the treatment (Day 141) will be 20 weeks.
  Interventions: Drug: Semaglutide
- Placebo (Semaglutide) (Placebo Comparator): Participants will receive placebo (semaglutide). The treatment period from first treatment (Day 1) to end of the treatment (Day 141) will be 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Participants will receive gradually increasing doses of semaglutide (subcutaneous [s.c.], in the thigh, abdomen or upper arm) injection once weekly, until they reach a dose of level of 2.4 mg, which they will continue for 5 weeks.
  Arms: Semaglutide
Drug: Placebo — Participants will receive once weekly injections of semaglutide matched placebo.
  Arms: Placebo (Semaglutide)

SUMMARY:
This study will look at how the emptying of the participant's stomach after a meal is affected by semaglutide (a new medicine) compared to a "dummy" medicine. In addition, the study will also look at the effect of semaglutide on the participant's appetite and energy intake. Participants will either get semaglutide or "dummy" medicine - which treatment any participant gets is decided by chance. Participants will take 1 injection per week. The study medicine is injected with a thin needle in the stomach, thigh or upper arm. The study will last for about 27 weeks (from first treatment to last check-up). Participants will have 8 visits at the clinic with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 to 65 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 30.0 and 45.0 kg/m^2 (both inclusive)

Exclusion criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, or endocrinological conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
AUC0-5h,para: the area under the paracetamol concentration-time curve from 0 to 5 hours at steady state | 0 to 5 hours after standardised meal (day 142)
  Measured in h*micrograms/mL

SECONDARY OUTCOMES:
AUC0-1h,para: the area under the paracetamol concentration-time curve from 0 to 1 hour at steady state | 0 to 1 hour after standardised meal (day 142)
  Measured in h*micrograms/mL
Cmax,para: the maximum observed paracetamol concentration from 0 to 5 hours | 0 to 5 hours after standardised meal (day 142)
  Measured in micrograms/mL
Tmax,para: the time of maximum observed paracetamol concentration from 0 to 5 hours | 0 to 5 hours after standardised meal (day 142)
  Measured in hours
Energy intake during ad libitum lunch | Day 142
  Measured in kilojoules
Mean postprandial rating - Hunger (AUC30-300min/270 min) using visual analogue scales (VAS) from 30 up to 300 minutes during standardised breakfast meal | Day 142
  Measured in mm, from 0-100. The ends of each line indicate the most extreme sensation respondents have experienced.
Mean postprandial rating - Fullness (AUC30-300min/270 min) using VAS from 30 up to 300 minutes during standardised breakfast meal | Day 142
  Measured in mm, from 0-100. The ends of each line indicate the most extreme sensation respondents have experienced.
Mean postprandial rating - Satiety (AUC30-300min/270 min) using VAS from 30 up to 300 minutes during standardised breakfast meal | Day 142
  Measured in mm, from 0-100. The ends of each line indicate the most extreme sensation respondents have experienced.
Mean postprandial rating - Prospective food consumption (AUC30-300min/270 min) using VAS from 30 up to 300 minutes during standardised breakfast meal | Day 142
  Measured in mm, from 0-100. The ends of each line indicate the most extreme sensation respondents have experienced.
Mean postprandial rating - Overall appetite score (OAS) (AUC30-300min/270 min) using VAS from 30 up to 300 minutes during standardised breakfast meal | Day 142
  Measured in mm, from 0-100. The ends of each line indicate the most extreme sensation respondents have experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Friedrichsen M, Breitschaft A, Tadayon S, Wizert A, Skovgaard D. The effect of semaglutide 2.4 mg once weekly on energy intake, appetite, control of eating, and gastric emptying in adults with obesity. Diabetes Obes Metab. 2021 Mar;23(3):754-762. doi: 10.1111/dom.14280. Epub 2021 Jan 3. PMID 33269530